CLINICAL TRIAL: NCT02574845
Title: The Effect of Different Doses of Metformin or Furosemide on Rosuvastatin Pharmacokinetics Following Oral Administration in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Six-way Crossover Study)
Brief Title: DDI (Effect of Metformin and Furosemide on Rosuvastatin PK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 352.2094; 2015-003052-46 (EudraCT Number)
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Metformin; Furosemide

ARMS (6):
- R (Reference) Rosuvastatin (Experimental): 1film-coated tablet as single dose, fasted
  Interventions: Drug: Rosuvastatin
- T1 (Test 1) Rosuvastatin + Metformin HCl (Experimental): Rosuvastatin: 1 film-coated tablet as single dose (10 mg), fasted / Metformin HCl (10 mg) as single dose, fasted
  Interventions: Drug: Rosuvastatin; Drug: Metformin HCl
- T2 (Test 2) Rosuvastatin + Metformin HCl (Experimental): Rosuvastatin: 1 film-coated tablet as single dose (10 mg), fasted / Metformin HCl (50 mg) as single dose, fasted
  Interventions: Drug: Rosuvastatin; Drug: Metformin HCl
- T3 (Test 3) Rosuvastatin + Metformin HCl (Experimental): Rosuvastatin: 1 film-coated tablet as single dose (10 mg), fasted / Metformin HCl (500 mg) as single dose, fasted
  Interventions: Drug: Rosuvastatin; Drug: Metformin HCl
- T4 (Test 4) Rosuvastatin + Furosemide (Experimental): Rosuvastatin: 1 film-coated tablet as single dose (10 mg), fasted / Furosemide: (1 mg) as single dose, fasted
  Interventions: Drug: Rosuvastatin; Drug: Furosemide
- T5 (Test 5) Rosuvastatin + Furosemide (Experimental): Rosuvastatin: 1 film-coated tablet as single dose (10 mg), fasted / Furosemide: (5 mg) as single dose, fasted
  Interventions: Drug: Rosuvastatin; Drug: Furosemide

INTERVENTIONS:
Drug: Rosuvastatin
Drug: Metformin HCl
  Arms: T1 (Test 1) Rosuvastatin + Metformin HCl; T2 (Test 2) Rosuvastatin + Metformin HCl; T3 (Test 3) Rosuvastatin + Metformin HCl
Drug: Furosemide
  Arms: T4 (Test 4) Rosuvastatin + Furosemide; T5 (Test 5) Rosuvastatin + Furosemide

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of rosuvastatin when given alone (Reference treatment, R) compared to when given together with one of the three different doses of metformin (10 mg, Test treatment 1 (T1); 50 mg (T2); 500 mg (T3)) or one of the two doses of furosemide (1 mg (T4); 5 mg (T5)).

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
2. Age of 18 to 55 years (incl.)
3. BMI of 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts
9. Chronic or relevant acute infections
10. History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
11. Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
12. Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial
13. Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
14. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
15. Inability to refrain from smoking on specified trial days
16. Alcohol abuse (consumption of more than 30 g per day)
17. Drug abuse or positive drug screening
18. Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
19. Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
20. Inability to comply with dietary regimen of trial site
21. Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

    In addition, the following trial-specific exclusion criteria apply:
22. Myopathy
23. Hereditary galactose or fructose intolerance, lactase deficiency, or glucose-galactose malabsorption
24. Allergy or hypersensitivity against sulfonamides

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2015-12-09 (Actual); Study Completion 2015-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Stopfer P, Giessmann T, Hohl K, Sharma A, Ishiguro N, Taub ME, Jungnik A, Gansser D, Ebner T, Muller F. Effects of Metformin and Furosemide on Rosuvastatin Pharmacokinetics in Healthy Volunteers: Implications for Their Use as Probe Drugs in a Transporter Cocktail. Eur J Drug Metab Pharmacokinet. 2018 Feb;43(1):69-80. doi: 10.1007/s13318-017-0427-9. PMID 28685495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were screened for eligibility to participate in the study. No run-in or wash-out period was conducted, since the trial was conducted in healthy subjects, that were not expected to take medications regularly. Actual number of subjects enrolled in fact represents randomized subjects due to the study set up.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that they (the subjects) met all strictly implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- Treatment (T) 1-T3-Reference (REF)-T5-T2-T4: The subjects received test treatment 1 (T1) which is 10 milligram (mg) metformin hydrochloride (oral solution, brand name: MetfoLiquid GeriaSan) together with the reference treatment (REF) which is rosuvastatin (film-coated, brand name: Crestor) followed by test treatment 3 (T3) which is 500mg metformin hydrochloride together with REF followed by REF alone followed by test treatment 5 (T5) which is 5 mg furosemide (oral solution, brand name: Lasix liquidum) together with REF followed by test treatment 2 (T2) which is 50 mg of metformin hydrochloride together with REF followed by test treatment 4 (T4) which is 1mg of furosemide together with REF. Trial medication was administered as a single oral dose in the fasted state in each treatment period. The six single dose treatment periods were separated from each other by a wash-out period of at least 6 days between the drug administrations.
- T2-REF-T4-T1-T5-T3: The subjects received T2, followed by REF alone, followed by T4, followed by T1, followed by T5 and followed by T3. Trial medication was administered as a single oral dose in the fasted state in each treatment period. The six single dose treatment periods were separated from each other by a wash-out period of at least 6 days between the drug administrations.
- T3-T5-T1-T4-REF-T2: The subjects received T3, followed by T5, followed by T1, followed by T4, followed by REF alone and followed by T2. Trial medication was administered as a single oral dose in the fasted state in each treatment period. The six single dose treatment periods were separated from each other by a wash-out period of at least 6 days between the drug administrations.
- T4-T2-T5-REF-T3-T1: The subjects received T4, followed by T2, followed by T5, followed by REF alone, followed by T3 and followed by T1. Trial medication was administered as a single oral dose in the fasted state in each treatment period. The six single dose treatment periods were separated from each other by a wash-out period of at least 6 days between the drug administrations.
- T5-T4-T3-T2-T1-REF: The subjects received T5, followed by T4, followed by T3, followed by T2, followed by T1 and followed by REF alone. Trial medication was administered as a single oral dose in the fasted state in each treatment period. The six single dose treatment periods were separated from each other by a wash-out period of at least 6 days between the drug administrations.
- REF-T1-T2-T3-T4-T5: The subjects received REF alone, followed by T1, followed by T2, followed by T3, followed by T4 and followed by T5. Trial medication was administered as a single oral dose in the fasted state in each treatment period. The six single dose treatment periods were separated from each other by a wash-out period of at least 6 days between the drug administrations.
Period: Overall Study
Arm/Group | Treatment (T) 1-T3-Reference (REF)-T5-T2-T4 | T2-REF-T4-T1-T5-T3 | T3-T5-T1-T4-REF-T2 | T4-T2-T5-REF-T3-T1 | T5-T4-T3-T2-T1-REF | REF-T1-T2-T3-T4-T5
Started | 3 | 3 | 3 | 3 | 3 | 3
Received T1 | 3 | 2 | 3 | 3 | 2 | 2 (one subject missed treatment period 2)
Received T2 | 3 | 3 | 3 | 3 | 2 | 3
Received T3 | 2 (one subject missed treatment period 2) | 2 | 3 | 3 | 2 | 3
Received T4 | 3 | 2 | 3 | 3 | 2 | 2
Received T5 | 3 | 2 | 3 | 3 | 3 | 2
Received R | 3 | 2 | 3 | 3 | 2 | 3
Completed | 3 | 2 | 3 | 3 | 2 | 2
Not Completed | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Consent withdrawn further participation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomised set (RS) includes all randomised subjects, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (T) 1-T3-Reference (REF)-T5-T2-T4 | T2-REF-T4-T1-T5-T3 | T3-T5-T1-T4-REF-T2 | T4-T2-T5-REF-T3-T1 | T5-T4-T3-T2-T1-REF | REF-T1-T2-T3-T4-T5 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (2.6) | 33.0 (8.7) | 39.3 (10.3) | 32.0 (14.1) | 22.0 (2.6) | 37.3 (12.9) | 31.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Rosuvastatin From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: This outcome measure presents the area under the concentration-time curve of rosuvastatin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: Blood sampling within 3 hours (h) prior to the study drug administration, at the time of administration (0:00) and 30 minutes, 1h, 1:30h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 11h, 12h, 24h, 34h, and 48h thereafter.
Population: The pharmacokinetic (PK) parameter set (PKS) includes all randomised subjects who took at least one dose of study medication and provided at least one primary or secondary PK parameter that was not excluded from analysis due to non-evaluability or protocol violation relevant for the evaluation of the pharmacokinetics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol) * hour (h) / Litre (L)
Groups:
- REF Alone: The subjects received the reference treatment (REF) which is rosuvastatin (film-coated, brand name: Crestor). Trial medication was administered as a single oral dose in the fasted state.
- Treatment 1: The subjects received test treatment 1 which is 10 mg metformin hydrochloride (oral solution, brand name: MetfoLiquid GeriaSan) together with the reference treatment (REF) which is rosuvastatin (film-coated, brand name: Crestor). Trial medication was administered as a single oral dose in the fasted state.
- Treatment 2: The subjects received test treatment 2 which is 50 mg metformin hydrochloride (oral solution, brand name: MetfoLiquid GeriaSan) together with the reference treatment (REF) which is rosuvastatin (film-coated, brand name: Crestor). Trial medication was administered as a single oral dose in the fasted state.
- Treatment 3: The subjects received test treatment 3 which is 500 mg metformin hydrochloride (oral solution, brand name: MetfoLiquid GeriaSan) together with the reference treatment (REF) which is rosuvastatin (film-coated, brand name: Crestor). Trial medication was administered as a single oral dose in the fasted state.
- Treatment 4: The subjects received test treatment 4 which is 1 mg furosemide (oral solution, brand name: Lasix liquidum) together with the reference treatment (REF) which is rosuvastatin (film-coated, brand name: Crestor). Trial medication was administered as a single oral dose in the fasted state.
- Treatment 5: The subjects received test treatment 5 which is 5 mg furosemide (oral solution, brand name: Lasix liquidum) together with the reference treatment (REF) which is rosuvastatin (film-coated, brand name: Crestor). Trial medication was administered as a single oral dose in the fasted state.
Arm/Group | REF Alone | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 16 | 15 | 16 | 15 | 15 | 16
nanomol (nmol) * hour (h) / Litre (L) | 81.5 (50.9) | 87.8 (54.5) | 88.7 (62.4) | 126 (66.7) | 91.5 (55.4) | 97.2 (52.7)
Statistical Analysis 1: Comparison: REF Alone vs Treatment 1; This statistical analysis assess the effect of coadministration of 10 mg metformin hydrochloride on the primary outcome measure of the REF treatment; Test type: Superiority or Other; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including the effects: 'sequence', 'subjects within sequence', 'period' and 'treatment'; Adjusted geometric mean ratio T1/REF (%) = 101.95, 90% CI 2-sided [89.49 to 116.15]
Statistical Analysis 2: Comparison: REF Alone vs Treatment 2; This statistical analysis assess the effect of coadministration of 50 mg metformin hydrochloride on the primary outcome measure of the REF treatment; Test type: Superiority or Other; ANOVA; ANOVA model on the logarithmic scale including the effects: 'sequence', 'subjects within sequence', 'period' and 'treatment'; Adjusted geometric mean ratio T2/REF (%) = 106.09, 90% CI 2-sided [96.12 to 117.11]
Statistical Analysis 3: Comparison: REF Alone vs Treatment 3; This statistical analysis assess the effect of coadministration of 500 mg metformin hydrochloride on the primary outcome measure of the REF treatment; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T3/REF (%) = 152.18, 90% CI 2-sided [135.12 to 171.41]
Statistical Analysis 4: Comparison: REF Alone vs Treatment 4; This statistical analysis assess the effect of coadministration of 1 mg furosemide on the primary outcome measure of the REF treatment; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T4/REF (%) = 106.97, 90% CI 2-sided [94.34 to 121.30]
Statistical Analysis 5: Comparison: REF Alone vs Treatment 5; This statistical analysis assess the effect of coadministration of 5 mg furosemide on the primary outcome measure of the REF treatment; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T5/REF (%) = 115.92, 90% CI 2-sided [101.93 to 131.82]

2. Primary Outcome: Maximum Concentration of Rosuvastatin (Cmax)
Description: This outcome measure presents the maximum measured concentration of rosuvastatin in plasma (Cmax).
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | REF Alone | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 16 | 15 | 16 | 15 | 15 | 16
nmol/L | 9.04 (52.4) | 9.59 (60.5) | 9.94 (69.4) | 14.0 (71.2) | 9.90 (62.0) | 10.8 (62.7)
Statistical Analysis 1: Comparison: REF Alone vs Treatment 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T1/REF (%) = 102.47, 90% CI 2-sided [87.19 to 120.42]
Statistical Analysis 2: Comparison: REF Alone vs Treatment 2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T2/REF (%) = 106.98, 90% CI 2-sided [92.54 to 123.69]
Statistical Analysis 3: Comparison: REF Alone vs Treatment 3; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T3/REF (%) = 154.07, 90% CI 2-sided [131.70 to 180.24]
Statistical Analysis 4: Comparison: REF Alone vs Treatment 4; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T4/REF (%) = 106.81, 90% CI 2-sided [91.78 to 124.30]
Statistical Analysis 5: Comparison: REF Alone vs Treatment 5; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T5/REF (%) = 117.98, 90% CI 2-sided [98.27 to 141.65]

3. Secondary Outcome: Area Under the Curve of Rosuvastatin From 0 Extrapolated to Infinity (AUC0-∞)
Description: This outcome measure presents area under the concentration-time curve of rosuvastatin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | REF Alone | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Number analyzed (Participants) | 15 | 14 | 16 | 14 | 15 | 16
nmol*h/L | 99.7 (39.0) | 105 (48.0) | 102 (55.0) | 149 (49.8) | 108 (47.9) | 115 (42.0)
Statistical Analysis 1: Comparison: REF Alone vs Treatment 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T1/REF (%) = 101.22, 90% CI 2-sided [89.23 to 114.82]
Statistical Analysis 2: Comparison: REF Alone vs Treatment 2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T2/REF (%) = 107.26, 90% CI 2-sided [97.65 to 117.81]
Statistical Analysis 3: Comparison: REF Alone vs Treatment 3; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T3/REF (%) = 146.45, 90% CI 2-sided [135.21 to 158.62]
Statistical Analysis 4: Comparison: REF Alone vs Treatment 4; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T4/REF (%) = 105.63, 90% CI 2-sided [92.20 to 121.00]
Statistical Analysis 5: Comparison: REF Alone vs Treatment 5; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 2]; Adjusted geometric mean ratio T5/REF (%) = 118.10, 90% CI 2-sided [106.75 to 130.67]

ADVERSE EVENTS:
Time Frame: From the first administration of study medication to the end of the 4 day residual effect period (96 hours after each administration of study medication) up to 24 days in total.
Arm/Group | REF Alone | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Treatment 5
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/17 | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 4/15 | 2/17 | 2/15 | 3/15 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | REF Alone (N=16) | Treatment 1 (N=15) | Treatment 2 (N=17) | Treatment 3 (N=15) | Treatment 4 (N=15) | Treatment 5 (N=16)
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes